CLINICAL TRIAL: NCT03644186
Title: Phase II Open-label, Multicentre, Randomized Trial of Neoadjuvant Palbociclib in Combination With Hormonal Therapy and HER2 Blockade Versus Paclitaxel in Combination With HER2 Blockade for Postmenopausal Patients With Hormone Receptor Positive/HER2 Positive Early Breast Cancer
Brief Title: To Reduce the Use of Chemotherapy in Postmenopausal Patients With ER-positive and HER2-positive Breast Cancer (TOUCH)
Acronym: TOUCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Pfizer (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 55-17; 2017-005067-40 (EudraCT Number)
Record Dates: First submitted 2018-08-14; First posted 2018-08-23 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Estrogen Receptor Positive Tumor; HER2-positive Breast Cancer
Keywords: hormone receptor positive early breast cancer; HER2 receptor positive early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab; pertuzumab; palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel plus trastuzumab and pertuzumab (Active Comparator): Receiving paclitaxel 80mg/m2 i.v. on day 1, 8, 15 every 28 days for 4 cycles, trastuzumab 600mg s.c. every 3 weeks for a total of 5 doses and pertuzumab 840 mg i.v. loading dose followed by 420 mg i.v. every 3 weeks for a total of 5 doses.
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab
- Palbociclib plus letrozole plus trastuzumab and pertuzumab (Experimental): Receiving palbociclib 125 mg/day orally for 21 days followed by 7 day's rest, for four 28 day cycles, letrozole 2.5 mg/day orally for 16 weeks and trastuzumab 600 mg s.c. every 3 weeks for a total of 5 doses and pertuzumab 840 mg i.v. loading dose followed by 420 mg i.v. every 3 weeks for 5 doses.
  Interventions: Drug: Palbociclib; Drug: Letrozole; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Paclitaxel — Chemotherapy plus HER2 Blockade
  Other Names: Paclitaxel Sandoz
  Arms: Paclitaxel plus trastuzumab and pertuzumab
Drug: Trastuzumab — Chemotherapy plus HER2 Blockade
  Other Names: Herceptin
  Arms: Paclitaxel plus trastuzumab and pertuzumab
Drug: Pertuzumab — Chemotherapy plus HER2 Blockade
  Other Names: Perjeta
  Arms: Paclitaxel plus trastuzumab and pertuzumab
Drug: Palbociclib — CDK Inhibition plus Hormonal Therapy plus HER2 Blockade
  Other Names: Ibrance
  Arms: Palbociclib plus letrozole plus trastuzumab and pertuzumab
Drug: Letrozole — CDK Inhibition plus Hormonal Therapy plus HER2 Blockade
  Other Names: Femara
  Arms: Palbociclib plus letrozole plus trastuzumab and pertuzumab
Drug: Trastuzumab — CDK Inhibition plus Hormonal Therapy plus HER2 Blockade
  Other Names: Herceptin
  Arms: Palbociclib plus letrozole plus trastuzumab and pertuzumab
Drug: Pertuzumab — CDK Inhibition plus Hormonal Therapy plus HER2 Blockade
  Other Names: Perjeta
  Arms: Palbociclib plus letrozole plus trastuzumab and pertuzumab

SUMMARY:
This is a phase II open-label, multicentre, randomized trial. The study assesses the treatment of postmenopausal patients with hormone receptor positive/HER2 positive early breast cancer with neoadjuvant palbociclib in combination with hormonal therapy and HER2 blockade, versus the treatment with paclitaxel in combination with HER2 blockade.

DETAILED DESCRIPTION:
TOUCH is an open label, international, phase II neoadjuvant trial which will assess the treatment of elderly patients with hormone receptor positive / human epidermal growth factor receptor-2 (HER2) positive early breast cancer with neoadjuvant palbociclib in combination with hormonal therapy and HER2 blockade, versus the treatment with paclitaxel in combination with HER2 blockade.

The neo-adjuvant setting was chosen to evaluate these therapy combinations in a short time-frame and to provide access to biomaterial both at baseline and after the end of the treatment, at surgery. Biopsy specimens will be analyzed at the end of the trial by gene-expression profiling to assess RBsig status. This marker may represent a tool to identify the participants who are more likely to benefit from a chemotherapy-free regimen in this population.

Palbociclib is a potent, highly selective, reversible, orally active, inhibitor of cyclin-dependent kinases 4 and 6 (CDK 4/6), therefore inhibiting cell growth and can be safely and effectively administered to older patients without need for dose adjustment based solely on age. Treatment de-escalation, namely harnessing and taking maximum advantage of targeted therapies vs conventional treatment (chemotherapy) in order to limit side effects, is particularly appealing in the older population.

Clinical data from the HR positive /HER2 negative setting show that combinations of palbociclib and letrozole are safe and effective. These combinations have not yet been tested in the HR positive /HER2 positive population that the investigators include in this trial. However, combinations of trastuzumab and endocrine treatment (ET), including letrozole have shown to be safe and to have some additional activity compared to ET alone in the HR positive /HER2 positive population. Therefore, the role of palbociclib in addition to letrozole and trastuzumab plus pertuzumab needs to be further studied.

Current standard of care for treatment of HER2 positive BC incorporates chemotherapy and anti-HER2 agents, with chemotherapy regimens of sequential anthracyclines and taxanes, used as single agents or in combination with other chemotherapy drugs. Trastuzumab is often administered concurrently with a single agent taxane to avoid the possible additive cardiac toxicity of combinations of anthracycline containing regimens and trastuzumab.

A regimen of weekly paclitaxel and trastuzumab plus pertuzumab was chosen as the comparator arm in this trial. More aggressive chemotherapy may not be justified in this population and trial participants may receive additional treatment after surgery, at the discretion of the treating doctor.

Preclinical and clinical rationale exists to support the proposal that palbociclib may represent a valuable option for increasing the activity of ET and anti-HER2 agents, such that a triple combination with these agents could prove superior to a standard treatment with chemotherapy and anti-HER2 agents.

The investigators hypothesize that the combination of palbociclib, letrozole and trastuzumab plus pertuzumab proposed in this trial will be more efficacious compared to the combinations of anti-HER2 agents and ET reported in other trials.

In 2019, it is estimated that of 260,600 newly diagnosed cases of invasive breast cancer in the United States, 82% occurred in women aged 50 or over. Furthermore, of the 41,760 breast cancer-related deaths in the same year, 90% occurred in this predominantly post-menopausal age group. Around 40% of BCs occur in women aged 65 and older. Of these, 10-15% have tumors that overexpress HER2. Elderly patients are generally underrepresented in clinical trials and may benefit from anti-HER2 agents as much as the younger population. Post-menopausal patients with HR positive /HER2 positive BC represent a unique group of patients with an unmet clinical need. This population is the focus of the TOUCH trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer, with the following characteristics:

   * Early breast cancer with tumor size >1 cm (as measured by at least one of the required examination methods of clinical examination, mammography and ultrasonography);
   * No clinical evidence of regional lymph node metastasis (via physical and/or radiological exam) (cN0) OR
   * Clinical evidence of cN1 status, defined by nodal involvement limited to clinically or radiologically detectable metastasis to movable ipsilateral level I, II axillary lymph node(s)
   * No evidence of metastasis (M0).
2. Postmenopausal, defined by women with:

   * Prior bilateral surgical oophorectomy; OR
   * Amenorrhea and age ≥60 years; OR
   * Age <60 years and amenorrhea for 12 or more consecutive months in the absence of alternative pathological or physiological cause (including chemotherapy, tamoxifen, toremifene, ovarian suppression, or hormonally-based contraception) plus FSH and serum estradiol levels within the laboratory's reference ranges for postmenopausal women
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Primary tumor must have positive estrogen receptor (ER) ≥10%
5. Primary tumor must be HER2-positive (by IHC and/or ISH)
6. Baseline LVEF ≥55% measured by Echocardiography (preferred) or MUGA scan
7. Normal hematologic status:

   * Absolute neutrophil count ≥1500/mm3 (1.5 × 109/L);
   * Platelets ≥100 × 109/L;
   * Hemoglobin ≥9 g/dL (≥90 g/L).
8. Normal renal function: serum creatinine ≤1.5 ULN
9. Normal liver function:

   * Serum total bilirubin ≤1.5 × upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (<2 × ULN) is allowed;
   * AST or ALT ≤2.5 × ULN;
   * Alkaline phosphatase ≤2.5 × ULN.
10. Written Informed Consent (IC) must be signed and dated by the patient and the Investigator prior to randomization.
11. The patient has been informed of and agrees to data transfer and handling, in accordance with national data protection guidelines.
12. The patient agrees in writing to make tumor (mandatory diagnostic core biopsy and surgical specimen) available for submission for central pathology review and to conduct translational studies as part of this protocol.

Exclusion Criteria:

1. Tumor of any size with direct extension to the chest wall and/or to the skin (ulceration or skin nodules) (T4 according to AJCC 8th edition cancer staging TNM)
2. Inflammatory breast cancer
3. Bilateral invasive breast cancer
4. Received any prior treatment for primary invasive breast cancer
5. Any active tumor of non-breast-cancer histology
6. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina pectoris, ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (NYHA functional classification ≥II), cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
7. Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety
8. Contraindications or known hypersensitivity to any of the trial medications or excipients
9. Treatment with any investigational agents within 30 days prior to expected start of trial treatment
10. Any GI disorder that may affect absorption of oral medications, such as malabsorption syndrome or status post major bowel resection
11. Evidence via physical and/or radiological exam of cN2 or cN3 nodal involvement defined by: metastasis to ipsilateral level I, II axillary lymph nodes that are clinically fixed or matted, OR involvement of ipsilateral infraclavicular, internal mammary and/or supraclavicular lymph node(s)
12. History of extensive disseminated/bilateral or known presence of interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and pulmonary fibrosis. A history of prior radiation pneumonitis is not considered an exclusion criterion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Biganzoli, MD, Study Chair — USL4 Hospital of Prato, Italy; Etienne Brain, MD, Study Chair — Institut Curie, Paris, France
Locations (54):
- Belgium (6):
  - AZ Klina, Augustijinslei 100, Brasschaat
  - Jules Bordet Institute, Brussels
  - CHR de la Citadelle, Boulevard du XIIe de Ligne, 1, Liège
  - Clinique Saint- Joseph, Rue de Hesbaye 75, Liège
  - Clinique Saint Elizabeth, Place Louise Godin 15, Namur
  - AZ Nikolaas, Moerlandstrat 1, Sint-Niklaas
- France (15):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Léon Berard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Institut de Cancérologie de l'Ouest (ICO), Nantes
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Institut Curie - Site de Paris, Paris
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Site Saint Cloud, Saint-Cloud
  - Clinique Pasteur, Toulouse
  - Institut Claudius Regaud, Toulouse
- Italy (22):
  - Clinica Oncologica-Ospedali Riuniti Ancona, Via Conca n.71,, Torrette, Ancona
  - Istituto scientifico Romagnolo per lo studio e la cura,Via Piero Maroncelli 40, Meldola, Forli
  - U.O Medicina Oncologica Ospedale di Carpi, Via G. Molinari, 2, Carpi, Modena
  - Centro di Riferimento Oncologico (CRO), Via Franco Gallini 2, Aviano, Pordenone
  - ASO "SS Antonio e Biagio Cesare Arrigo, Via Venezia 16, Alessandria
  - Ospedali Riuniti di Bergamo, A.O.Papa Giovanni XXIII, Piazza OMS1, Bergamo
  - Ospedale S. Orsola-Malpighi, Viale Ercolani 4/2, Bologna
  - Comprensorio Sanitario Bolzano, Via Lorenz Bohler, 5, Bolzano
  - ASST Spedali Civili Brescia, Piazzale Spedali Civili n.1, Brescia
  - E.O. Ospedali Galliera, Mura delle Cappuccine, 14, Genova
  - Ospedale Policlinico San Martino,Largo Rosanna Benzi,10, Genova
  - Ospedale Civile di Lecco,Via della Filanda 14, Lecco
  - Milano, IEO, Via Ripamonti 435, Milan
  - Università del Piemonte Orientale - SCDU Oncologia, Corso Mazzini 18, Novara
  - Azienda Ospedaliero-Universitaria di Parma, via Gramsci 14, Parma
  - Istituti Clinici Scientifici Maugeri SpA-SB,Via Salvatore Maugeri N° 10, Pavia
  - A.O. Universitaria Pisana Ospedale Santa Chiara Pisa, Via Roma 67, Pisa
  - Hospital of Prato, Via Dolce dei Mazzamuti, 7, Prato
  - Santa Maria delle Croci Hospital, Viale Randi 5, Ravenna
  - UO Oncologia, Rimini Hospital, Via Settembrini 2, Rimini
  - Azienda Ospedaliero-Universitaria di Udine, Piazzale S.M. Misericordia 15, Udine
  - AO Universitaria Ospedale Di Circolo e Fondazione,v.le L. Borri, 57, Varese
- Switzerland (11):
  - Kantonsspital Baden AG, Baden, Aarau
  - Universitatsspital Basel, Petersgraben 4, Basel, Canton of Basel-City
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - University Hospital Zurich, Frauenklinikstrasse 10, Zurich, Canton of Zurich
  - Oncology Institute of Southern Switzerland (IOSI), Ospedale San Giovanni, IOSI, Bellinzona, Canton Ticino
  - Brustzentrum Thurgau / Kantonsspital Frauenfeld, Pfaffenholzstrasse 4, Frauenfeld, Thurgau
  - Inselspital Bern, Bern
  - HFR Freiburg - Kantonsspital, Fribourg
  - University Hospital Geneva, Geneva
  - Kantonsspital St. Gallen, Rorschacher Strasse 95, Sankt Gallen
  - Brust-Zentrum AG, Seefeldstrasse 214, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biganzoli L, Wildiers H, Oakman C, Marotti L, Loibl S, Kunkler I, Reed M, Ciatto S, Voogd AC, Brain E, Cutuli B, Terret C, Gosney M, Aapro M, Audisio R. Management of elderly patients with breast cancer: updated recommendations of the International Society of Geriatric Oncology (SIOG) and European Society of Breast Cancer Specialists (EUSOMA). Lancet Oncol. 2012 Apr;13(4):e148-60. doi: 10.1016/S1470-2045(11)70383-7. Epub 2012 Mar 30. PMID 22469125
- [Background] Biganzoli L, Aapro M, Loibl S, Wildiers H, Brain E. Taxanes in the treatment of breast cancer: Have we better defined their role in older patients? A position paper from a SIOG Task Force. Cancer Treat Rev. 2016 Feb;43:19-26. doi: 10.1016/j.ctrv.2015.11.009. Epub 2015 Dec 15. PMID 26827689
- [Background] Cancer Genome Atlas Network. Comprehensive molecular portraits of human breast tumours. Nature. 2012 Oct 4;490(7418):61-70. doi: 10.1038/nature11412. Epub 2012 Sep 23. PMID 23000897
- [Background] Cristofanilli M, Turner NC, Bondarenko I, Ro J, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Zhang K, Theall KP, Jiang Y, Bartlett CH, Koehler M, Slamon D. Fulvestrant plus palbociclib versus fulvestrant plus placebo for treatment of hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3): final analysis of the multicentre, double-blind, phase 3 randomised controlled trial. Lancet Oncol. 2016 Apr;17(4):425-439. doi: 10.1016/S1470-2045(15)00613-0. Epub 2016 Mar 3. PMID 26947331
- [Background] Demidenko E. Sample size and optimal design for logistic regression with binary interaction. Stat Med. 2008 Jan 15;27(1):36-46. doi: 10.1002/sim.2980. PMID 17634969
- [Background] Finn RS, Dering J, Conklin D, Kalous O, Cohen DJ, Desai AJ, Ginther C, Atefi M, Chen I, Fowst C, Los G, Slamon DJ. PD 0332991, a selective cyclin D kinase 4/6 inhibitor, preferentially inhibits proliferation of luminal estrogen receptor-positive human breast cancer cell lines in vitro. Breast Cancer Res. 2009;11(5):R77. doi: 10.1186/bcr2419. PMID 19874578
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Herschkowitz JI, He X, Fan C, Perou CM. The functional loss of the retinoblastoma tumour suppressor is a common event in basal-like and luminal B breast carcinomas. Breast Cancer Res. 2008;10(5):R75. doi: 10.1186/bcr2142. Epub 2008 Sep 9. PMID 18782450
- [Background] Jenkins EO, Deal AM, Anders CK, Prat A, Perou CM, Carey LA, Muss HB. Age-specific changes in intrinsic breast cancer subtypes: a focus on older women. Oncologist. 2014 Oct;19(10):1076-83. doi: 10.1634/theoncologist.2014-0184. Epub 2014 Aug 20. PMID 25142841
- [Background] Johnston S, Pippen J Jr, Pivot X, Lichinitser M, Sadeghi S, Dieras V, Gomez HL, Romieu G, Manikhas A, Kennedy MJ, Press MF, Maltzman J, Florance A, O'Rourke L, Oliva C, Stein S, Pegram M. Lapatinib combined with letrozole versus letrozole and placebo as first-line therapy for postmenopausal hormone receptor-positive metastatic breast cancer. J Clin Oncol. 2009 Nov 20;27(33):5538-46. doi: 10.1200/JCO.2009.23.3734. Epub 2009 Sep 28. PMID 19786658
- [Background] Kaufman B, Mackey JR, Clemens MR, Bapsy PP, Vaid A, Wardley A, Tjulandin S, Jahn M, Lehle M, Feyereislova A, Revil C, Jones A. Trastuzumab plus anastrozole versus anastrozole alone for the treatment of postmenopausal women with human epidermal growth factor receptor 2-positive, hormone receptor-positive metastatic breast cancer: results from the randomized phase III TAnDEM study. J Clin Oncol. 2009 Nov 20;27(33):5529-37. doi: 10.1200/JCO.2008.20.6847. Epub 2009 Sep 28. PMID 19786670
- [Background] Malorni L, Piazza S, Ciani Y, Guarducci C, Bonechi M, Biagioni C, Hart CD, Verardo R, Di Leo A, Migliaccio I. A gene expression signature of retinoblastoma loss-of-function is a predictive biomarker of resistance to palbociclib in breast cancer cell lines and is prognostic in patients with ER positive early breast cancer. Oncotarget. 2016 Sep 13;7(42):68012-68022. doi: 10.18632/oncotarget.12010. PMID 27634906
- [Background] Miles D, Baselga J, Amadori D, Sunpaweravong P, Semiglazov V, Knott A, Clark E, Ross G, Swain SM. Treatment of older patients with HER2-positive metastatic breast cancer with pertuzumab, trastuzumab, and docetaxel: subgroup analyses from a randomized, double-blind, placebo-controlled phase III trial (CLEOPATRA). Breast Cancer Res Treat. 2013 Nov;142(1):89-99. doi: 10.1007/s10549-013-2710-z. Epub 2013 Oct 16. PMID 24129974
- [Background] Witkiewicz AK, Ertel A, McFalls J, Valsecchi ME, Schwartz G, Knudsen ES. RB-pathway disruption is associated with improved response to neoadjuvant chemotherapy in breast cancer. Clin Cancer Res. 2012 Sep 15;18(18):5110-22. doi: 10.1158/1078-0432.CCR-12-0903. Epub 2012 Jul 18. PMID 22811582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The TOUCH study was activated on 4 October 2018. The first patient was enrolled on 16 April 2019. The protocol was updated (18 February 2020) to relax the eligibility criteria in order to increase the accrual rate; expanded from women greater than or equal to 65 to postmenopausal patients. The last patient was enrolled on 28 July 2022. The final accrual was 147 patients (target 144) in 37 centers in 4 countries. Out of 147 randomized patients 2 patients did not start any protocol treatment.
Period: Overall Study
Arm/Group | Paclitaxel Plus Trastuzumab and Pertuzumab | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab
Started | 74 | 73
Completed | 73 | 72
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The TOUCH study was activated on 4 October 2018. The first patient was enrolled on 16 April 2019. The protocol was updated (18 February 2020) to relax the eligibility criteria in order to increase the accrual rate; expanded from women greater than or equal to 65 to postmenopausal patients. The last patient was enrolled on 28 July 2022. The final accrual was 147 patients (target 144) in 37 centers in 4 countries. Out of 147 randomized patients 2 patients did not start any protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel Plus Trastuzumab and Pertuzumab | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab | Total
Number analyzed (Participants) | 74 | 73 | 147
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 21 | 23 | 44
  >=65 years | 53 | 50 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 10 | 11 | 21
  Italy | 44 | 41 | 85
  France | 7 | 6 | 13
  Switzerland | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR)
Description: Pathological complete response (pCR) is defined as absence of invasive tumour cells in the breast and in the axillary lymph nodes at the time of surgery (ypT0/ypTis ypN0) determined from the local histopathologic evaluation according to the American Joint Committee on Cancer Staging Manual. The presence of in situ cancer after trial treatment in the absence of residual invasive disease constitutes a pCR.
Time Frame: Assessed within 30 days of the time of breast surgery after completion of a treatment period of up to 16 weeks; up to 21 weeks. If the patient does not undergo surgery, assessment will occur within 30 days after all treatment is stopped; up to 30 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Plus Trastuzumab and Pertuzumab | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab
Number analyzed (Participants) | 73 | 72
Participants | 24 | 24

2. Secondary Outcome: Pathological Complete Response (pCR) in the Breast
Description: Defined as the absence of invasive tumour cells in the breast at the time of surgery (ypT0/ypTis) determined from the local histopathologic evaluation according to the American Joint Committee on Cancer Staging Manual..
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Plus Trastuzumab and Pertuzumab | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab
Number analyzed (Participants) | 73 | 72
Participants | 26 | 25

3. Secondary Outcome: Objective Response
Description: The number of patients with partial or complete response measured physically by caliper and by ultrasound and mammography. Response was assessed using World Health Organization tumor measurement and response criteria.
  Complete response (CR) - The disappearance of all known disease. Partial response (PR) - A 50% or more decrease in total tumor size, i.e., the sum of the products of the maximal diameter (MD) and the corresponding largest perpendicular diameter (LPD) of the lesions which have been measured to determine the effect of therapy. In addition, there can be no appearance of new lesions or progression of any lesion.
  Stable disease (SD) - Neither a 50% decrease in total tumor size, nor a 25% increase in the size of one or more measurable lesions has been determined.
  Progressive disease (PD) - An increase of least 25% in total tumor size relative to the smallest size measured during the trial.
Time Frame: Tumor assessments were performed by ultrasound and mammography at screening (prior to treatment start), and before surgery; measurements by caliper were assessed at the same time points and at the end of cycle 2 (28 days/cycle), approximately 56 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Plus Trastuzumab and Pertuzumab | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab
Number analyzed (Participants) | 73 | 72
Participants
  Objective response - complete response | 35 | 38
  Objective response - partial response | 17 | 19
  Objective response - stable disease | 4 | 4
  Objective response - progressive disease | 3 | 2
  Objective response - not evaluable | 14 | 9

4. Secondary Outcome: Rate of Breast Conserving Surgery (BCS)
Description: Defined as the number of patients undergoing BCS, divided by the number of patients in the assessable population (subset of the randomized population with RBsig status successfully determined who received at least 1 dose of medication).
Time Frame: From randomization until completion of study, up to 20 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Plus Trastuzumab and Pertuzumab | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab
Number analyzed (Participants) | 73 | 72
Participants | 49 | 59

ADVERSE EVENTS:
Time Frame: Assessed at the end of every 4-week cycle until the end of trial treatment prior to surgery; up to 20 weeks. Only serious adverse events were assessed 30 days after end of treatment; up to 21 weeks.
Description: The severity and causality will be classified according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5. The CTCAE is available for downloading on the internet at http://evs.nci.nih.gov/ftp1/CTCAE/About.html. For this trial, Grade 1s were not collected for non-targeted adverse events and hence are not included in the reporting of Other (not including serious) adverse event table.
Arm/Group | Paclitaxel Plus Trastuzumab and Pertuzumab | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/72
Serious Adverse Events (participants affected / at risk) | 23/73 | 39/72
Other Adverse Events (participants affected / at risk) | 68/73 | 69/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel Plus Trastuzumab and Pertuzumab (N=73) | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab (N=72)
Neutrophil count decreased (Investigations) | 5 | 31
Diarrhea (Gastrointestinal disorders) | 8 | 6
Infections (Infections and infestations) | 0 | 2
Skin and cutaneous disorders (Skin and subcutaneous tissue disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 4
Ejection fraction decreased (Infections and infestations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 — Cystoid macular edema
Fatigue (General disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Ileal obstruction (Gastrointestinal disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel Plus Trastuzumab and Pertuzumab (N=73) | Palbociclib Plus Letrozole Plus Trastuzumab and Pertuzumab (N=72)
Neutrophil count decreased (Investigations) | 12 | 23
Anemia (Blood and lymphatic system disorders) | 36 | 35
Platelet count decreased (Investigations) | 2 | 28
Nausea (Gastrointestinal disorders) | 19 | 16
Diarrhea (Gastrointestinal disorders) | 45 | 47
Thromboembolic event (Vascular disorders) | 2 | 1
Infections (Infections and infestations) | 18 | 14
Skin and cutaneous disorders (Skin and subcutaneous tissue disorders) | 30 | 22
Hypertension (Vascular disorders) | 7 | 1
Ejection fraction decreased (Investigations) | 4 | 2
Hepatobiliary disorder (Hepatobiliary disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 4
Stomach pain (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 8 | 2
Allergic reaction (Immune system disorders) | 8 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 1 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 0
Depression (Psychiatric disorders) | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Phlebitis (Vascular disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal mucositis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Conjunctivitis (Investigations) | 0 | 1
GGT increased (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0
Hot flashes (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol Part 1 (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03644186/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol Part 2 (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03644186/Prot_SAP_001.pdf